CLINICAL TRIAL: NCT02518581
Title: Estimating Free-living Human Energy Expenditure - Validation of the Doubly Labelled Water Method in Subjects With Type 2 Diabetes Mellitus
Brief Title: Validation of the Doubly Labelled Water Method in Subjects With Type 2 Diabetes Mellitus
Acronym: DLW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OBDM-03
Record Dates: First submitted 2015-08-03; First posted 2015-08-10 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doubly labelled water (Other)
  Interventions: Procedure: Doubly labelled water method

INTERVENTIONS:
Procedure: Doubly labelled water method — DLW (doubly labeled water) method measures isotope dilution spaces and elimination rates to assess total energy expenditure (TEE). After enriching the body water of a subject with DLW (2H and 18O), it is only necessary to collect urine samples at defined time points, usually over a period of 1-2 weeks, so that the measurement can be done in individuals able to engage in their typical habits without restrictions. The resulting TEE measurement represents an integral value over the measurement period.

SUMMARY:
The present study is an exploratory trial to establish a feasible DLW (doubly labelled water) protocol for implementation in clinical trials conducted at Profil Institut für Stoffwechselforschung, investigating treatment options for overweight and obesity in populations with and without diabetic comorbidity. The study aims at the practical validation of a 1-2-week DLW protocol in overweight and obese type 2 diabetic subjects.

Total Energy Expenditure (TEE) values as assessed by DLW will then be compared to (1) TEE as calculated based on individual anthropometric measurements (including body composition) using the Müller formula and the AEE (activity related energy expenditure) based on reported work place and leisure time activities and (2) TEE as calculated from measured REE (resting energy expenditure) as assessed by indirect calorimetry and the AEE based on information recorded by the subjects in a physical activity diary and corresponding pedometer counts. Moreover, TEE assessments will be repeated once (separated by 2-4 weeks) to determine intra-subject variability / re-test reliability of the measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained before any trial-related activities.
2. Stable weight +/- 5% for at least 3 months prior screening visit.
3. Male or female subject, 18-64 years of age, both inclusive.
4. Body Mass Index (BMI) >= 25 kg/m2.
5. Type 2 diabetes mellitus (as diagnosed clinically) ≥ 12 months.
6. HbA1c <= 9 % at screening visit.
7. Stable treatment (>= 3 month) with

   * Oral antidiabetics (OADs) (except OADs that are associated with a reduction in body weight (α-glucosidase inhibitors, sodium glucose transporter 2-inhibitors (SGLT2))) and/or
   * basal insulin injections and/or
   * a dietary regimen. Subjects on a basal-bolus insulin regimen will not be enrolled.
8. Considered generally healthy (apart from type 2 diabetes mellitus and with the exception of conditions associated with diabetes mellitus or the metabolic syndrome, such as dyslipidaemia and hypertension) upon completion of medical history, physical examination, vital signs, and analysis of laboratory safety variables, as judged by the Investigator.

Exclusion Criteria:

1. Clinical significant acute illness within 2 weeks before study procedures, including severe infections, as judged by the Investigator.
2. Receipt of any investigational medicinal product within 3 months before trial related procedures.
3. Mental incapacity or language barriers which preclude adequate understanding or cooperation, unwillingness to participate in the trial, known or suspected not to comply with study directives or not to be reliable or trustworthy, or subjects who in the opinion of their general practitioner or the Investigator should not participate in the trial.
4. Use of diuretics.
5. Intake of any other drug or dietary supplement that in the opinion of the Investigator may impair validity of energy expenditure assessments.
6. Clinically significant abnormal biochemistry screening tests, as judged by the Investigator. In particular, elevated liver enzymes (AST or ALT > 3 times the upper limit of normal) or impaired renal function with an estimated Glomerular Filtration Rate (eGFR; estimate after CKD-EP) < 60 ml/min.
7. Clinically significant abnormal electrocardiogram (ECG) findings at screening, as judged by the Investigator.
8. Positive alcohol breath test at screening visit.
9. Significant history of alcoholism or drug abuse as judged by the Investigator or consuming more than 21 units of alcohol per week (one unit of alcohol equals about 330 ml of beer, one glass of wine of 120 ml, or 40 ml spirits).
10. Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day) who is not able or willing to refrain from smoking and use of nicotine substitute products during the study.
11. Excessive consumption of coffee and tea (i.e. more than 5 cups/day), chocolate or beverages such as cola containing methylxanthine (caffeine, theophylline or theobromine) as judged by the investigator.
12. Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures include surgical sterilisation, hormonal intrauterine devices (coil), oral hormonal contraceptives, sexual abstinence or a surgically sterilised partner).
13. Type 1 diabetes mellitus, diabetes resulting from pancreatic injury, or secondary forms of diabetes, e.g., acromegaly or Cushing's syndrome.
14. History of hyperosmolar crisis, diabetic coma, or severe hypoglycemia within the last 3 months prior to trial examinations.
15. Use of weight-loss medication or any non-permitted antidiabetic medication that is associated with a reduction in body weight (α-glucosidase inhibitors, SGLT2-inhibitors) within 3 months before trial examination.
16. Use of injectable anti-diabetic therapy (other than insulin), e.g. GLP-1 receptor agonists (glucagon-like peptide), within 3 months prior to screening.
17. Steroid therapy other than topical application.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Free-living total energy expenditure | up to 3 month
  Assessed by doubly labelled water
Resting energy expenditure | up to 3 month
  Assessed by indirect calorimetry
Activity-induced energy expenditure | up to 3 month
  Assessed by diary and pedometer

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany